CLINICAL TRIAL: NCT02057796
Title: Systematic Empirical vs. Test-guided Anti-tuberculosis Treatment Impact in Severely Immunosuppressed HIV-infected Adults Initiating Antiretroviral Therapy With CD4 Cell Counts <100/mm3: the STATIS Randomized Controlled Trial
Brief Title: Systematic Empirical vs. Test-guided Anti-TB Treatment Impact in Severely Immunosuppressed HIV-infected Adults Initiating ART With CD4 Cell Counts <100/mm3
Acronym: STATIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12290
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; Tuberculosis; Systematic empiric TB treatment; ART; TB diagnosis; Xpert MTB/RIF®; Urine LAM
MeSH Terms: conditions — Tuberculosis | interventions — Diagnostic Imaging; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz; lamivudine, zidovudine drug combination; Rifampin; Isoniazid; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xpert MTB/RIF®, Determine TB LAM, Chest X-ray (Experimental): Arm1 Extensive TB screening:
  In this arm, point-of-care tests for TB will be used at randomization (in all patients) and at each scheduled or unscheduled follow-up visit (in patients with signs or symptoms suggestive of TB and no clear alternative diagnosis); TB treatment will only be prescribed to patients with a diagnosis of TB
  Interventions: Device: Xpert MTB/RIF®, Determine TB LAM, Chest X-ray; Drug: ART (Atripla, Truvada, Efavirenz, Combivir); Drug: Rifampin, isoniazid, pyrazinamide, ethambutol
- Rifampin, isoniazid, pyrazinamide, ethambutol (Experimental): Arm 2: Systematic Empiric treatment (Rifampicin,isoniazid, pyrazinamide, ethambutol) ART
  In this arm, all patients will start a systematic 6-month TB treatment at randomization. TB screening tests will not systematically be used neither at randomization nor while patients are on TB treatment.
  Interventions: Drug: ART (Atripla, Truvada, Efavirenz, Combivir); Drug: Rifampin, isoniazid, pyrazinamide, ethambutol

INTERVENTIONS:
Device: Xpert MTB/RIF®, Determine TB LAM, Chest X-ray — The following point-of-care TB tests will be systematically performed:
  Xpert MTB/RIF® on sputum (in all patients able to provide sputum; no sputum induction will be requested in others), Urine LAM (all patients). Depending on clinical presentation, Xpert MTB/RIF® will also be performed on any relevant extra-pulmonary specimen.
  TB treatment will depend on the result of the tests:
  Criteria met for confirmed or probable TB : TB treatment will be initiated immediately (Visit 1) followed by ART initiation 2 weeks later (Visit 2); No evidence of confirmed or probable TB: ART will be started immediately (Visit 1).
  Arms: Xpert MTB/RIF®, Determine TB LAM, Chest X-ray
Drug: ART (Atripla, Truvada, Efavirenz, Combivir) — * ART (TDF-3TC/FTC or AZT-3TC + efavirenz) will be started immediately after randomization in patients not put on TB treatment, and 2 weeks after initiation of TB treatment in others.
  * ART will be initiated 2 weeks after the onset of TB treatment (V2) for Arm 2
  Other Names: ART
Drug: Rifampin, isoniazid, pyrazinamide, ethambutol — Arm 1: Only patients who meet standardized criteria for TB at inclusion or during follow-up will receive a standard TB treatment (2ERHZ/4RH); Arm 2: • All patients will start a 6-month standard TB treatment (2ERHZ/4RH) at randomization
  Other Names: Systematic Empiric treatment

SUMMARY:
In countries with a high tuberculosis (TB) prevalence, TB and invasive bacterial infections are leading causes of early death in patients who initiate antiretroviral therapy (ART) with advanced immunodeficiency.

We hypothesize that a systematic 6-month empirical TB treatment initiated 2 weeks before the introduction of ART in HIV-infected adults with severe immunosuppression (CD4<100/mm3) and no overt evidence of TB will reduce the risk of death and invasive bacterial infections. This strategy will be compared to one of extensive TB testing using point-of-care tests (Xpert MTB/RIF® and urine lipoarabinomanan LAM) and chest X-ray to identify and treat only patients with at least one positive test suggestive of TB.

DETAILED DESCRIPTION:
Settings: Cambodia, Côte d'Ivoire, Uganda, Vietnam. Design: Multicentre, two-arm, unblinded randomized controlled superiority trial.

Objective: To compare the 24-week risk of death and occurrence of invasive bacterial infection between two experimental strategies in HIV-1 infected adults who start ART with a CD4 count <100/mm3: (i) continuous extensive TB screening during follow-up each time the patient present with symptoms, versus (ii) systematic empirical TB treatment started 2 weeks before ART initiation.

Trial strategies:

At inclusion, participants will be randomized 1:1 in two strategies of TB testing and treatment: extensive TB screening, or systematic empirical TB treatment.

Extensive TB screening (arm 1): In this arm:

* TB screening point-of-care tests (Xpert MTB/RIF®, urine LAM) and chest X-ray will be used extensively at randomisation (in all patients) and during follow-up (in patients with signs or symptoms suggestive of TB);
* Only patients who meet standardized criteria for TB at inclusion or during follow-up will receive a standard TB treatment (2ERHZ/4RH);
* ART (tenofovir(TDF)-lamivudine (3TC)/emtricitabine(FTC) or zidovudine (AZT)-lamivudine+ efavirenz) will be started immediately after randomization in patients not put on TB treatment, and 2 weeks after initiation of TB treatment in others.

Systematic empirical TB treatment (arm 2): In this arm:

* TB screening point-of-care tests will not be used;
* All patients will start a 6-month standard TB treatment (2ERHZ/4RH) at randomization; ART (tenofovir-lamivudine/emtricitabine or zidovudine-lamivudine+ efavirenz) will be started 2 weeks after TB treatment initiation.

Both strategies will apply to the first 24 weeks in the trial (intervention period).

From week-24 to week-48, the choice of TB tests and the prescription of TB treatment will be left upon the decision of the investigator in both trial arms.

Inclusion time: 24 months. Follow-up: each patient will be followed 48 weeks. Statistical analysis: the primary analysis will be intention to treat. It will compare the 24-week probability of death or invasive bacterial infection between arms.

Sample size: 1050 participants. This will allow demonstration of a 40% reduction in the 24-week probability of death or invasive bacterial infection in arm 2, compared to arm 1 (α 5%; 1-β 80%).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* HIV-1 infection as documented at any time prior to trial entry, as per national testing procedures;
* CD4 <100 cells/mm3;
* No history of antiretroviral drug use (except transient ART for PMTCT);
* Able to correctly understand the trial and to sign the informed consent.

Exclusion Criteria:

* HIV-2 co-infection;
* Contra-indication to efavirenz;
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >5 times the upper limit of normal;
* Creatinine clearance <50 ml/min;
* Overt evidence that TB treatment should be started immediately;
* History of TB treatment in the past 5 years;
* Ongoing TB chemoprophylaxis (isoniazid preventive therapy);
* Any condition that would lead to differ ART initiation (e.g. acute condition requiring investigations and/or treatment prior to ART initiation);
* Current pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
All-cause mortality and incidence of invasive bacterial infections | 24 weeks
  The primary endpoint is the composite of (i) 24-week all-cause mortality and (ii) 24-week incidence of invasive bacterial infections

SECONDARY OUTCOMES:
Incidence of confirmed/probable/possible TB | 24 Weeks and 48 weeks
Incidence of grade 3 or 4 adverse events | 24 Weeks and 48 weeks

OTHER OUTCOMES:
Incidence of TB-associated IRIS | 24 Weeks and 48 Weeks
Incidence of AIDS-defining diseases other than TB | 24 Weeks and 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier Blanc, MD, PhD, Principal Investigator — Université de Nantes, Institut du thorax, CHU Nantes, France; Kouao Médard Serge Domoua, MD, Principal Investigator — Service de Pneumologie, CHU de Treichville, Abidjan, Côte d'Ivoire
Locations (4):
- Sihanouk Hospital Center of Hope, Phnom Penh, Cambodia
- CePReF Centre de Prise en charge de Recherche et de Formation, Abidjan, Yopougon, Côte d’Ivoire
- ISS ImmunoSuppression Service, Mbarara, Uganda
- Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Bonnet M, Gabillard D, Domoua S, Muzoora C, Messou E, Sovannarith S, Nguyen DB, Badje A, Juchet S, Bunnet D, Borand L, Natukunda N, Tran TH, Anglaret X, Laureillard D, Blanc FX; Systematic empirical vs. Test-guided Anti-tuberculosis Treatment Impact in Severely immunosuppressed HIV-infected adults initiating antiretroviral therapy with CD4 cell counts <100/mm3 (STATIS) Agence Nationale de Recherche sur le Sida et les hepatites virales (ANRS) 12290 Trial Team. High Performance of Systematic Combined Urine Liboarabinomannan Test and Sputum Xpert MTB/RIF for Tuberculosis Screening in Severely Immunosuppressed Ambulatory Adults With Human Immunodeficiency Virus. Clin Infect Dis. 2023 Jul 5;77(1):112-119. doi: 10.1093/cid/ciad125. PMID 36883573
- [Derived] Blanc FX, Badje AD, Bonnet M, Gabillard D, Messou E, Muzoora C, Samreth S, Nguyen BD, Borand L, Domergue A, Rapoud D, Natukunda N, Thai S, Juchet S, Eholie SP, Lawn SD, Domoua SK, Anglaret X, Laureillard D; STATIS ANRS 12290 Trial Team. Systematic or Test-Guided Treatment for Tuberculosis in HIV-Infected Adults. N Engl J Med. 2020 Jun 18;382(25):2397-2410. doi: 10.1056/NEJMoa1910708. PMID 32558469

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02057796/SAP_000.pdf